CLINICAL TRIAL: NCT05567354
Title: A Randomized, Double-blind, Placebo-and Active-Controlled Crossover Study to Evaluate the Intranasal Abuse Potential of PF614 Compared with Immediate-Release Oxycodone and Placebo in Non-Dependent Recreational Opioid Users
Brief Title: A Study to Evaluate the Intranasal Abuse Potential of PF614 in Non-Dependent Recreational Opioid Users (PF614-103)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ensysce Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PF614-103
Record Dates: First submitted 2022-05-22; First posted 2022-10-05 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2022-12

CONDITIONS: Recreational Drug Use
MeSH Terms: conditions — Recreational Drug Use | interventions — Oxycodone; Tablets

STUDY DESIGN:
Intervention Model Description: This will be a 3 way crossover study to evaluate the abuse potential of PF614.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind treatment and randomization will be used to reduce potential bias during data collection and evaluation of clinical endpoints. A placebo control will be used to establish the frequency and magnitude of changes in clinical endpoints that may occur in the absence of active treatment, as well as to minimize subject and investigator bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- PF614 100 mg capsule (Experimental): Eligible subjects will be admitted to the clinical site on Day-1. Subjects will receive PF614 100mg capsules in a randomized, double-blind, crossover manner.
  Interventions: Drug: PF614
- Oxycodone HCl tablets (Active Comparator): Eligible subjects will be admitted to the clinical site on Day -1. Subjects will receive crushed oxycodone HCl IR 40mg in a randomized, double-blind, crossover manner.
  Interventions: Drug: Oxycodone
- Placebo powder in capsules (Placebo Comparator): Eligible subjects will be admitted to the clinical site on Day-1. Subjects will receive Placebo powder in a randomized, double-blind, crossover manner.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PF614 — PF614 100 mg capsules
  Other Names: Oxycodone prodrug
  Arms: PF614 100 mg capsule
Drug: Oxycodone — Oxycodone HCl IR 40mg
  Other Names: Oxycodone hydrochloride (HCl) immediate-release (IR) tablets
  Arms: Oxycodone HCl tablets
Other: Placebo — placebo powder
  Arms: Placebo powder in capsules

SUMMARY:
The purpose of this study is to examine the abuse potential and pharmacokinetics of PF614 compared with a non-abuse deterrent, commercially available, immediate release (IR) oxycodone hydrochloride (HCl) formulation and placebo.

DETAILED DESCRIPTION:
This will be a randomized, double-blind, placebo-and active-controlled, 3-way crossover study to evaluate the abuse potential and pharmacokinetics of intranasally administered PF614, relative to crushed oxycodone HCl IR tablets and placebo in non-dependent recreational opioid users. The study will consist of 4 phases: Screening, Qualification, Treatment, and Follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, aged 18 to 55 years, inclusive, in good general health.
2. Body mass index (BMI) within the range of 18.0 to 33.0 kg/m2, inclusive, and a minimum weight of 50.0 kg.
3. Current opioid users who have used opioids for recreational (non-therapeutic) purposes (i.e., for psychoactive effects) at least 10 times in the past year and at least once in the 12 weeks before Screening.
4. Must have experience with intranasal opioids for the purpose of recreational (non-therapeutic) use on at least 3 occasions in the year prior to Screening.
5. Must not be physically dependent on opioids, as demonstrated by successful completion of the Naloxone Challenge Test.
6. Must meet Drug Discrimination Test eligibility criteria (Section 8.3).
7. Female subjects must have a negative serum pregnancy test at Screening and a negative urine pregnancy test at randomization. Post-menopausal women (i.e., no menstrual period for at least one year) must have a follicle-stimulation hormone (FSH) level >30 milli-international unit (mIU)/mL at Screening.
8. Female subjects must use a medically acceptable method of birth control (oral or transdermal contraceptives, condom, spermicidal foam, intrauterine device (IUD), progestin implant or injection, heterosexual abstinence, vaginal ring or sterilization of partner) from the time of Screening through 2 weeks after the last study treatment.
9. Male subjects must agree to use medically acceptable methods of contraception (diaphragm/sponge/condom with spermicide, vasectomy), and/or their female sexual partners of childbearing potential must be using and willing to continue to use medically acceptable contraception (i.e., hormonal oral contraceptive pills, patches, or vaginal rings, contraceptive implant or injection intrauterine contraceptive system [with or without hormone]) from Screening and for at least 90 days after the last study drug administration.
10. Able to speak, read and understand English sufficiently to allow completion of all study assessments.
11. Subjects must be able to provide meaningful written informed consent.
12. Subjects must be willing and able to follow study instructions and be likely to complete all study requirements.

Exclusion Criteria:

1. Substance or alcohol dependence (excluding nicotine and caffeine) within the past 2 years, as defined by the Diagnostic and Statistical Manual of Mental Disorders - Fourth Edition - Text Revision (DSM IV-TR), and/or has ever participated or plans to participate in a substance or alcohol rehabilitation program to treat their substance or alcohol dependence.
2. History or presence of clinically significant abnormality as assessed by physical examination, medical history, electrocardiograms (ECGs), vital signs or laboratory values, which, in the opinion of the investigator, would jeopardize the safety of the subject or the validity of the study results. Retesting may be permitted at the discretion of the investigator.
3. History or presence of acute respiratory depression, chronic pulmonary disease, cor pulmonale, delirium tremens, central nervous system (CNS) depression, or increased cerebrospinal or intracranial pressure.
4. Documented history of or currently active seizure disorder (excluding febrile seizures in childhood) or history of clinically significant head injury or syncope of unknown origin.
5. History of gastrointestinal disturbance requiring frequent use of antacids.
6. Subjects with a history of suicidal ideation within the past 6 months or a lifetime history of suicidal behavior, as assessed by the C SSRS (baseline version).
7. Heavy smoker (>20 cigarettes per day) and/or is unable to abstain from smoking while housed at the clinical site.
8. History of allergy or hypersensitivity to oxycodone, any other opioid or naloxone.
9. Female subjects who are currently pregnant (have a positive pregnancy test) or lactating or who are planning to become pregnant within 30 days of last study drug administration.
10. Positive for hepatitis B surface antigen (HBsAg), hepatitis C, human immunodeficiency virus (HIV) or severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
11. Evidence of clinically significant hepatic or renal impairment, including alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >1.5 × the upper limit of normal (ULN). Retesting may be permitted at the discretion of the investigator.
12. Donation or loss of more than 500 mL whole blood within 30 days preceding entry into the Treatment Phase.
13. Difficulty with venous access or unsuitable or unwilling to undergo catheter insertion.
14. Use of a prohibited medication or investigational product, as specified in Section 9.7.1.
15. Is an employee of the sponsor or research site personnel directly affiliated with this study, or is an immediate family member of any of these persons, defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
16. Falls under any other condition, that, in the investigator's opinion, (i) puts the subject at increased risk, (ii) could confound the study results, (iii) may interfere significantly with the subject's participation in the study, or (iv) has the potential to limit the subject's ability to complete the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Peak Maximum Effect (Emax) for Drug Liking (At this Moment) Visual Analog Scale (VAS) | Up to 24 hour post-dose (up to Day 2)
  Relative abuse potential of PF614 compared to Oxycodone and Placebo (I). Emax for drug liking VAS will be reported. Drug liking VAS is a bipolar scale designed to assess a participant's liking for a given study intervention at the time the question is being asked (that is, at this moment). It is scored as an integer ranging from 0 (strong disliking) to 100 (strong liking)
Take Drug again VAS (Emax) | 12 and 24 hours post-dose
  Relative abuse potential of PF614 compared to Oxycodone and Placebo (II). Emax for take drug again VAS will be reported. Peak effect for take drug again based on bipolar VAS from 0 (definitely no) to 100 (definitely so).

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | Up to 24 hour post-dose (up to Day 2)
  Compare the peak plasma concentration of oxycodone derived from PF614 and oxycodone derived from oxycodone IR tablets
Time to Peak Plasma Concentration (Tmax) | Up to 24 hour post-dose (up to Day 2)
  Compare the time to peak plasma concentration of oxycodone derived from PF614 and oxycodone derived from oxycodone IR tablets
Area Under the Curve Plasma Concentration (AUC 0-24) | Up to 24 hour post-dose (up to Day 2)
  Compare the 0-24 hr pharmacokinetic profile of oxycodone derived from PF614 and oxycodone derived from oxycodone IR tablets
Adverse events (AEs) | Through study completion, an average of 7 weeks
  Safety
Serious adverse events (SAEs) | Through study completion, an average of 7 weeks
  Safety
AEs leading to discontinuation | Through study completion, an average of 7 weeks
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: Glen Apseloff, MD, FCP, Principal Investigator — Ohio Clinical Trials
Locations (1):
- Ohio Clinical Trails, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirkpatrick DL, Evans C, Pestano LA, Millard J, Johnston M, Mick E, Schmidt WK. Clinical evaluation of PF614, a novel TAAP prodrug of oxycodone, versus OxyContin in a multi-ascending dose study with a bioequivalence arm in healthy volunteers. Clin Transl Sci. 2024 Mar;17(3):e13765. doi: 10.1111/cts.13765. PMID 38511523
- [Background] Kirkpatrick DL, Schmidt WK, Morales R, Cremin J, Seroogy J, Husfeld C, Jenkins T. In vitro and in vivo assessment of the abuse potential of PF614, a novel BIO-MD prodrug of oxycodone. J Opioid Manag. 2017 Jan/Feb;13(1):39-49. doi: 10.5055/jom.2017.0366. PMID 28345745